CLINICAL TRIAL: NCT03397186
Title: An Analysis of the Changes in the Sarcoma Tumor Immune Microenvironment Following Trabectedin
Brief Title: Immune Changes Following Trabectedin in Patients With Metastatic or Unresectable Sarcoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 9769; NCI-2017-02298 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9769 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG9217026 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-01-05; First posted 2018-01-11 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Myxoid Liposarcoma; Round Cell Liposarcoma; Stage III Soft Tissue Sarcoma AJCC v7; Stage IV Soft Tissue Sarcoma AJCC v7; Metastatic Soft Tissue Sarcoma; Unresectable Soft Tissue Sarcoma
MeSH Terms: conditions — Liposarcoma, Myxoid; Sarcoma | interventions — Biopsy; Trabectedin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Basic science (trabectedin, biopsy) (Other): Patients undergo a biopsy at baseline and then receive trabectedin for up to 4 cycles. Beginning 1 week after completion of cycle 2 and prior to cycle 3, patients undergo a second biopsy. Patients who achieve clinical benefit (CR, PR, SD) after the first post-treatment scan and who continue trabectedin for 4 cycles undergo a third biopsy after cycle 4.
  Interventions: Procedure: Biopsy; Other: Laboratory Biomarker Analysis; Drug: Trabectedin

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: Bx
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Trabectedin — Given as standard of care
  Other Names: Ecteinascidin; ecteinascidin 743; ET-743; Yondelis

SUMMARY:
This research trial studies the immune changes following trabectedin in patients with sarcoma that has spread to other places in the body (metastatic) or cannot be removed by surgery (unresectable). Analyzing tumor tissue may help to understand the changes in immune cells in or around the tumor or if there is an increase in immune cells in the tumor after receiving trabectedin.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Percentage of tumor tissue in pre- and post-treatment biopsies comprised of T-cells, as determined by flow cytometry.

SECONDARY OBJECTIVES:

I. To explore additional potential biomarkers including: numbers of tumor associated macrophage (TAM) in tumor II. To explore additional potential biomarkers including: phenotype (classically activated macrophages [M1] versus [vs] alternatively activated macrophages [M2]) as characterized by CD163, CD115, CD206 on infiltrating TAM.

III. To explore additional potential biomarkers including: phenotype of T cells infiltrating tumor (CD4, CD8, markers of CD4 phenotype including FoxP3 and memory).

IV. To explore additional potential biomarkers including: expression T cell inhibitory markers (PD-1, CTLA-4, TIM3).

V. To explore additional potential biomarkers including: recognition of autologous tumor by expanded tumor infiltrating lymphocyte lines.

VI. To explore additional potential biomarkers including: in tumor infiltrating lymphocyte (TIL) expanded from myxoid/round cell liposarcomas, recognition of cancer testis antigens.

OUTLINE:

Patients undergo a biopsy at baseline and then receive trabectedin for up to 4 cycles. Beginning 1 week after completion of cycle 2 and prior to cycle 3, patients undergo a second biopsy. Patients who achieve clinical benefit (complete response [CR], partial response [PR], stable disease [SD]) after the first post-treatment scan and who continue trabectedin for 4 cycles undergo a third biopsy after cycle 4.

After completion of study, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of advanced (unresectable or metastatic) sarcoma, for which trabectedin treatment is indicated
* Subjects must have received prior anthracycline treatment; subjects who failed to tolerate it or for whom it is not clinically appropriate in the opinion of their treating physician may be included
* All ongoing toxicities related to prior therapy must be resolved to grade 1 or better (except alopecia)
* Total bilirubin level =< upper limit of normal (ULN) mg/dL
* Aspartate aminotransferase (AST) =< 2.5 x ULN
* Alanine aminotransferase (ALT) =< 2.5 x ULN
* Alkaline phosphatase < 2.5 x ULN
* Serum creatinine =< 1.5 x ULN
* Calculated creatinine clearance >= 30 mL/min using the Cockcroft-Gault formula may be included
* Creatine phosphokinase (CPK) =< 2.5 x ULN
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelet count >= 100 x 10^9/L
* Hemoglobin >= 9 g/dL
* Baseline left ventricular ejection fraction (LVEF) 45% or greater (by echocardiogram or multigated acquisition scan [MUGA] study) and no evidence of New York Heart Association class ll to IV heart failure
* Subjects with lesions safely accessible for biopsy, in the opinion of the treating physician and/or interventional radiology
* Male or non-pregnant and non-breast feeding female:

  * Females of child-bearing potential must agree to use highly effective contraception without interruption from initiation of therapy and while on study medication and have a negative serum pregnancy test (beta-human chorionic gonadotropin [hCG]) result at screening and agree to ongoing pregnancy testing during the course of the study, and at the end of study treatment; a highly effective method of contraception is defined as one that results in a low failure rate (that is, < 1% per year), when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, or a vasectomized partner
  * Male subjects must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Ability to understand and sign informed consent
* Willingness and ability to comply with scheduled visits, laboratory tests, and other study procedures

Exclusion Criteria:

* Subjects for whom treatment with trabectedin is not indicated
* All subjects with brain metastases, except those meeting the following criteria:

  * Brain metastases that have been treated locally and are clinically stable for at least 2 weeks prior to enrollment
  * No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
  * Subjects must be either off steroids or on a stable or decreasing dose of =< 10 mg daily prednisone (or equivalent), excluding dexamethasone given as pre-treatment for trabectedin
* Prior organ transplantation, including allogeneic stem cell transplantation
* Subjects with abnormal prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) or bleeding diathesis
* Prior treatment with trabectedin
* Prior chemotherapy within 2 weeks; prior immunotherapy or biologic therapy within 4 weeks; prior radiation therapy within 3 weeks
* Significant acute or chronic infections as these may affect the immune response including:

  * Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
  * Positive test for hepatitis B virus (HBV) surface antigen and / or confirmatory hepatitis C virus (HCV) ribonucleic acid (RNA) (if anti-HCV antibody tested positive)
* Subjects on chronic therapy with any systemic immunosuppressant (not counting inhaled steroids or steroid creams) for any reason, including autoimmune disease
* Known alcohol or drug abuse
* Subjects who are breast feeding
* Subjects with known hypersensitivity including anaphylaxis to trabectedin
* Myocardial infarction (infarct) within 6 months before enrollment, New York Heart Association (NYHA) class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage change of T cells (CD3+) by flow cytometry | Baseline up to 4 weeks
  Analysis will be performed using a Wilcoxon matched-pairs assigned rank test as these will be paired samples where parametric distribution cannot be assumed. T cell receptor (TCR) sequencing, immunohistochemistry and gene expression analysis will all be used in order to confirm the primary endpoint.

SECONDARY OUTCOMES:
Expression of inhibitory ligands including PD-1, CTLA-4, LAG-3 on infiltrating T cells | Up to 4 weeks
  Gene expression will be analyzed using differential cluster analysis in order to look for patterns and gene groups that are differentially expressed in the post-treatment samples and such gene groups will be represented by heatmaps in order to illustrate this quantitative information. TCR fraction, clonality, and maximum (max) frequency will be compared between pre and post treatment samples.
CD8+ or CD4+ phenotype of infiltrating T cells | Up to 4 weeks
  Gene expression will be analyzed using differential cluster analysis in order to look for patterns and gene groups that are differentially expressed in the post-treatment samples and such gene groups will be represented by heatmaps in order to illustrate this quantitative information. TCR fraction, clonality, and max frequency will be compared between pre and post treatment samples.
Type 1 helper cell (Th1) versus (vs.) type 2 helper cell (Th2) phenotype of infiltrating T cells based on expression of CCR5 and CXCR3 | Up to 4 weeks
  Gene expression will be analyzed using differential cluster analysis in order to look for patterns and gene groups that are differentially expressed in the post-treatment samples and such gene groups will be represented by heatmaps in order to illustrate this quantitative information. TCR fraction, clonality, and max frequency will be compared between pre and post treatment samples.
Infiltrating tumor associated macrophage number | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seth Pollack, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No